CLINICAL TRIAL: NCT01462760
Title: Contribution of Actigraphy for the Evaluation of Elbow Range of Motion in the Joint Assessment in Gerontology
Acronym: BIOVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Principal Investigator, Del Cont Delphine, Professeur, Centre Hospitalier Universitaire de Nice
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-PP-11
Record Dates: First submitted 2011-10-12; First posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Geriatric Disorder
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First assessment: inclinometer (Other): First assessment: inclinometer Second assessment: actigraph and inclinometer
  Interventions: Device: Assessment with inclinometer
- first: Inclinometer and actigraph (Other): first: Inclinometer and actigraph second: inclinometer
  Interventions: Device: Assessment with inclinometer; Device: Assessment with actigraph

INTERVENTIONS:
Device: Assessment with inclinometer — joint assessment with inclinometer. The inclinometer used in this trial is Baseline® Bubble Inclinometer
Device: Assessment with actigraph — joint assessment with actigraph The actigraph used in this trial is the Motion Pod. It's an analysis and reeducation systems by biofeedback. The manufacturer is Movea.
  Arms: first: Inclinometer and actigraph

SUMMARY:
In this study, the investigators will measure range of motion of the elbow in a geriatric assessment in 85 subjects aged 65 years or over. These measures will be made by an actigraph and the software analysis BioVal. This technique will be compared with the standard technique (inclinometer). It will also be evaluated during this study, the ease of use and feedback.

DETAILED DESCRIPTION:
The deterioration of the musculoskeletal system occurring in aging is a major cause of loss of autonomy and directly affects the quality of life of the individual.

Support and appropriate rehabilitation for the patient's return home is essential. It requires physiotherapy assessment, which includes, among other things, a joint assessment with a measure passive range of motion.

Physical therapists have different techniques to achieve these measures for each of them, the benefits (time, reliability) and disadvantages. Among them, the goniometer and inclinometer are technical references The main objective of the study is to validate the MotionPod and the software BioVal as valid tool for measuring range of motion of the elbow in a joint geriatric assessment.

Secondary objectives are the study of the reproducibility of the measurement time and ease of use The measurement range of motion in the elbow in degree, estimated by actigraphy and software BioVal will be compared to those obtained with an inclinometer.

The movements are examined successively flexion, extension, pronation and supination.

The proportion of valid measurements will be calculated for each movement. The confidence interval 95% partner will also be calculated.

Moreover, in order to judge the validity of actigraphy in all of these measures, the investigators will calculate the proportion of patients for which the measures are valid for all four movements and the confidence interval 95% partner.

85 patients aged 65 years or more will be recruited at the Cimiez hospital the CHU of Nice, in the services of short, medium and long geriatric stay

ELIGIBILITY:
Inclusion Criteria:

* Prescription of physiotherapy .
* Prescription of a passive joint assessment
* Consent to participate in the study signed
* person with a social security system

Exclusion Criteria:

* person with a pacemeker
* patient with the inability to position the wrist straightness
* patient with the inability to position the shoulder in neutral
* metal prosthesis or osteosynthesis
* patient with a joint debate <20 °
* contraindicated warm up

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Inclinometer and actigraph assessment | elbow joint measures are done just at one time point, during the visit
  Elbow joint measures by the inclinometer and the actigraph

SECONDARY OUTCOMES:
Assessment of easily use | Assessment are done just at one time point, during the visit
  Assessment of easily use
Assessment comfort and utility of use | Assessment are done just at one time point, during the visit
  Assessment of comfort and utility of use
measurement time | Assessment are done just at one time point, during the visit
  measurement time

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Centre Memoire Ressources et Recherche, CHU de Nice, Nice, France

REFERENCES:
- [Derived] Sacco G, Turpin JM, Marteu A, Sakarovitch C, Teboul B, Boscher L, Brocker P, Robert P, Guerin O. Inertial sensors as measurement tools of elbow range of motion in gerontology. Clin Interv Aging. 2015 Feb 23;10:491-7. doi: 10.2147/CIA.S70452. eCollection 2015. PMID 25759568